CLINICAL TRIAL: NCT01469949
Title: Effect of Mental Imagery in Improvement of the Repositioning Accuracy and Proprioception in Patients With Low Back Pain
Brief Title: Mental Imagery Enhances Proprioception in Patients With Low Back Pain
Acronym: MI
Status: Completed | Type: Observational
Sponsor: Lebanese University (Other)
Responsible Party: Principal Investigator, Ahmad Rifai Sarraj, Head of Department of Physical Therapy, Lebanese University
Other Study IDs: LEBUNIV001
Record Dates: First submitted 2011-11-07; First posted 2011-11-10 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Low Back Pain
Keywords: Improvement of the accuracy of Lumbar repositioning
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Kinesthetic Imagery group: Subjects receiving Kinesthetic Imagery
  Interventions: Other: Watching or imagining movement
- Visual Imagery Group: Subjects receiving visual imagery
  Interventions: Other: Watching or imagining movement
- Control group: Subjects receiving measurement with intervention

INTERVENTIONS:
Other: Watching or imagining movement — Mental imagery are administered in two forms : kinesthetic when subjects imagine the movement of flexion and extension of the lumbar spine and Visual when subjects watch a video of a third person doing the flexion and extension movement
  Groups: Kinesthetic Imagery group; Visual Imagery Group

SUMMARY:
Mental imagery has been used in a variety of pathological instances in support to classical therapeutic treatments. The aim of the present study was to observe the effect of internal Kinesthetic and external Visual Imagery to improve proprioceptive feedback in low back pain. Fifty-five subjects with a history of low back pain were included in two experimental groups who used mental imagery and one control group who did not. The results showed the effectiveness of the Internal Kinesthetic Imagery to improve the accuracy of repositioning of lumbo-sacral spine that may subsequently improve the quality of the proprioceptive input. The possibility to use effectively mental imagery, as a part of proprioceptive rehabilitation process, is the principal outcome of this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suffering from common non-specific low back pain

Exclusion Criteria:

* Recent history of inner ear infection causing associated balance or coordination problems
* History of cerebral trauma followed by unresolved neurosensory symptoms
* Recent history of vestibular disorder and previous spinal surgery
* An involvement in specific balance or stabilization training during the 6 months prior testing. Patients taking pain medication were excluded from the study.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Fifty-five patients, with a history of common low back pain, have participated to the study. The subjects have been randomly distributed in two experimental groups and one control group. The gender, age, weight and height characteristics of the three groups (Visual Imagery Group, VIG; Kinesthetic Imagery Group, KIG; and Control Group, CG) are presented in Table 1. The patients presented no history of neurological or psychiatric disease, and gave their informed written consent.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of Lumbar Spine Repositioning | 2hours
  Before and after the intervention (Kinesthetic or visual Imagery)

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Physical Therapy, Beirut, Hadath, Lebanon